CLINICAL TRIAL: NCT05766228
Title: Web-Based Intercultural Given to Midwifery Students The Effect of Midwifery Education on Cultural Sensitivity and Cultural Skill Level
Brief Title: Web-Based Intercultural Midwifery Training Given to Midwifery Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kutahya Health Sciences University (Other)
Collaborators: Ataturk University (Other); Amasya University (Other); Çankırı Karatekin University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: E-15189967-050.02.04-145388
Record Dates: First submitted 2023-01-13; First posted 2023-03-13 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2023-01

CONDITIONS: Midwifery
Keywords: Web-Based Training; Intercultural Midwifery; Cultural Sensitivity; Cultural Skill

STUDY DESIGN:
Intervention Model Description: A Randomized Controlled, Multicenter Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Web-Based Intercultural Midwifery Training
  Interventions: Other: Web-Based Intercultural Midwifery Training
- Control (No Intervention): without any intervention

INTERVENTIONS:
Other: Web-Based Intercultural Midwifery Training — The training program is a program where students can log in via the internet using the password given to them by a smartphone or computer. The web base is compatible with mobile phones and is suitable for use at any time of the day. The trainings were prepared and explained by the researchers on the web page in the form of a video presentation with the theory-based didactic classroom technique using a Power Point presentation. The training program covered six weeks and consisted of two sessions of 30 minutes each week. In the first five weeks, general information on the development of intercultural midwifery and the main components of cultural competence models are explained. In the last week, training was completed with case presentations in the form of two sessions.
  Arms: Experimental

SUMMARY:
In this study, web-based intercultural midwifery training will increase students' cultural sensitivity and cultural skill level score averages. Based on these results, interactive training methods should be use on the web base to increase the effectiveness of the training given to the students and this training should be make widespread. It may be suggested that this research should be repeat using different training techniques and with different sample groups.

DETAILED DESCRIPTION:
International migrations have caused cultural diversity in societies (Foronda, 2008). Individuals from different societies have different needs due to habits from their cultures (Foronda, 2008; Henderson et al., 2018; Sharifi et al., 2019). Cultural diversity in countries has made the delivery of effective healthcare services difficult (Henderson et al., 2018). In this respect, the vaccination of the concepts of cultural competence and cultural sensitivity, which were popular in health service delivery, has become an international requirement for health professionals by coming to the fore in the literature (Henderson et al., 2018; Sharifi et al., 2019).

Lack of awareness about providing effective healthcare to patients from different cultures raises concerns about disrupting patient-clinician communication and causing inequality of access to care (Watt et al., 2016; Sharifi et al., 2019; Gungor et al., 2021). A society's values, beliefs, language characteristics, cultural structure, and living condition shape health promotion and protection behaviors (Henderson et al., 2018; Beser et al., 2021). On the other hand, providing culturally adequate and responsive care can be achieved by ensuring appropriate intercultural communication and approach competence (Çingöl et al., 2021). Health professionals who have cultural skills can act according to the rules and values of the society in which they provide health services, with high empathy skills, respect different cultures, and the most appropriate forms of communication with the culture (Mobula et al., 2015, Yılmaz et al., 2019).

The cultural or traditional practices are high in pregnancy, childbirth, and postpartum practices (Çakır Koçak & Sevil, 2015; Altuntuğ et al., 2018). The midwives should be sensitive to cultural differences to provide effective cultural care (Yılmaz et al., 2019; Guner et al., 2022). For this reason, it was necessary to integrate effective and appropriate cultural approaches to midwifery, which is closely related to women's health (Fleming et al., 2017; Beser et al., 2021; Gungor et al., 2021). At this point, it seems inevitable to prioritize the issues of raising awareness of cultural competence in midwifery education (Briscoe, 2013; Guner et al., 2022). The multicultural structure of Turkish society necessitates the informational support of midwives in understanding cultural differences, being sensitive, and meeting the needs of the society (Yılmaz et al., 2019; Guner et al., 2022). In the literature, to provide healthcare professionals with cultural competence and cultural sensitivity skills during undergraduate education were recommeded (Mobula et al., 2015; Yılmaz et al., 2019; Guner et al., 2022).

In a limited number of non-invasive studies on the subject, the focus was on defining the cultural competence and awareness of health professionals and students studying in the field of health (Aghajari et al., 2019; Shepherd et al., 2019; Beser et al., 2021; Çiftçi et al., 2021; Gungor et al., 2021). In some of the studies, the lack of interventional studies on increasing cultural skills was emphasized (Shepherd et al., 2019; Guner et al., 2022). In their study, Çingöl et al. (2021) reported that students' self-confidence and empathic skills increased in cultural sensitivity and intercultural communication as a result of an intercultural nursing course intervention. On the other hand, there is no interventional and multicenter study in the literature in which the cultural approaches of midwives and midwife candidates were developed. At this point, considering the prevalence of internet use worldwide (66.2%) (Internet World Stats, 2022), midwife candidates may gain cultural competencies through web-based training. The original results obtained from this study can contribute to the development of techniques that can be adapted to the cultural values of the societies where midwifery services are provided. Therefore, this study aims to examine the effect of web-based intercultural midwifery training given to students on students' cultural sensitivity and cultural skill level.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who agreed to participate in the study,
* who were between 18-25,
* who were midwifery students were included.

Exclusion Criteria:

* Students with any condition that hinders the research were not included.

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1113 (Actual)
Dates: Start 2022-10-15 (Actual); Primary Completion 2023-03-15 (Actual); Study Completion 2023-05-15 (Actual)

PRIMARY OUTCOMES:
Effect of web-based training | 12 weeks
  Measurement of cultural sensitivity and Measurement of Cultural Skill Level

CONTACTS AND LOCATIONS:
Locations (1):
- Kütahya Health Science University, Kütahya, Turkey (Türkiye)